CLINICAL TRIAL: NCT02058069
Title: Robotic Arm Assisted Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAKO Surgical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIOTKA_2014; 20131148 (Other: WIRB Protocol)
Record Dates: First submitted 2014-02-03; First posted 2014-02-07 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic Assisted Total Knee Arthroplasty (Experimental)
  Interventions: Device: Robotic Arm Assisted Total Knee Arthroplasty

INTERVENTIONS:
Device: Robotic Arm Assisted Total Knee Arthroplasty — The total knee implant system used for this study was the Kinetis implant system (MAKO Surgical Corp.).
  Other Names: MAKO Surgical Corp; RIO Total Knee Arthroplasty Application; MAKOplasty Total Knee Arthroplasty

SUMMARY:
The Investigation will be conducted as a single-submission, multi-center study with approval from and in compliance of the Western Institutional Review Board (WIRB).

The overall objective of this Investigation is to assess the safety and effectiveness of the Robotic Arm Interactive Orthopedic System (RIO) Total Knee Arthroplasty Application. Specifically, the study objectives are classified as follows:

* Primary Objective: Surgeon assessment of standardized TKA complications both intra-operatively and at short term follow up.
* Secondary Objective: Radiographic assessment of post-operative limb alignment.
* Supporting Objective: Patient assessment of post-operative function and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects may be recruited in to the Investigation.
* Age - The subject must be at least 21 years of age and skeletally mature as demonstrated radiographically by complete closure of the distal femoral and proximal tibial epiphyses.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigators and Approved Study Staff, are able to understand this Investigation and cooperate with the Investigation procedures and are willing to comply with all the required post-operative follow-ups.
* Subjects who require a total knee arthroplasty for primary surgical management of osteoarthritis, post-traumatic arthritis, rheumatoid arthritis, moderate deformities or femoral condyle osteonecrosis as defined below.
* Osteoarthritis: Kellgren-Lawrence Grade 3 or higher, with clinical history of an absence of major trauma to the joint; symptoms of pain, stiffness, swelling, and/or loss of motion; and with radiographic evidence of joint space narrowing, sub-chondral sclerosis, or peripheral osteophytes.
* Post-Traumatic Arthritis: Kellgren-Lawrence Grade 3 or higher, with a clinical history of trauma to the targeted knee and subsequent pain, stiffness, swelling and loss of motion; and with radiographic evidence of joint space narrowing, sub-chondral sclerosis, or peripheral osteophytes.
* Rheumatoid Arthritis: American College of Rheumatology classification score of 6 or higher, with a clinical history that demonstrates the following: morning stiffness for at least 1 hour and present for at least 6 weeks, swelling, loss of motion, and/or serum rheumatoid factor; and radiographic findings of narrow joint space, peri-articular osteopenia, and/or per-articular erosions.
* Moderate Deformities: Moderate varus, valgus, flexion, or post-traumatic deformities of no more than 15° assessed radiographically. Moderate recurvatum of no more than 8° assessed radiographically.
* Femoral Condyle Osteonecrosis: Loss of blood supply in the femoral condyle characterized by sudden onset of pain, possibly triggered by a specific seemingly routine activity or minor injury. Pain is often increased with activity and at night time and may cause swelling of the knee and sensitivity to touch and pressure and may result in limited motion. Confirmed by a bone scan, MRI, and/or x-ray.
* Subjects whose anatomy is appropriate for the available range of implant sizes.

Exclusion Criteria:

* Patients who have had previous surgical procedures requiring implantation of hardware in their operative side knee, hip, or ankle that would result in metal artifact scatter in a CT scan.
* Patients who have a fracture malunion of the distal femur or proximal tibia within 12cm of the knee center, assessed radiographically.
* Patients who are pregnant, may become pregnant during the course of the Investigation, or are currently lactating.
* Patients with allergies or suspected sensitivity to any patient-contacting component of the investigational device or the implant to be used in the study as listed below:
* Femoral component: Cobalt Chromium alloy (CoCr)
* Tibial component: Titanium alloy (Ti6Al4V)
* Tibial inserts and patella component: Vitamin E infused ultra-high molecular weight polyethylene (UHMWPE)
* Saw blade: 440C Stainless Steel
* Patients who require bilateral total knee arthroplasty.
* Patients who are currently on medical leave from their employment due to Workmen's Compensation.
* Patients who are currently state or federal prisoners.
* Patients who are currently Wards of the state.
* Patients who are at high risk for poor healing or confounding outcomes or at excessive risk for surgery i.e.: clinically significant/being actively treated for renal, hepatic, cardiac, hematologic, or neurologic disease or poorly controlled diabetes (HbA1c > 10 mg/dL) or previous history of joint infection.
* Patients who are known drug or alcohol abusers or with psychological disorders as defined by DSM V that could affect follow-up care or treatment outcomes.
* Patients who are currently involved in another clinical study with an investigational device.
* Patients with current litigation pending related to medical treatment of any sort.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Gustke, MD, Principal Investigator — Florida Orthopedic Institute, Tampa General Hospital; Thomas Coon, MD, Principal Investigator — Coon Joint Replacement Institute, St. Helena Hospital; Stefan Kreuzer, MD, Principal Investigator — Memorial Bone and Joint Research Foundation, Memorial Hermann Medical Center
Locations (3):
- United States (3):
  - Coon Joint Replacement Institue; St. Helena Hospital, St. Helena, California
  - Florida Orthopedic Institute, Tampa, Florida
  - Memorial Bone and Joint Research Foundation; Memorial Hermann Memorial City Medical Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Robotic Assisted Total Knee Arthroplasty: Participants who underwent primary total knee arthroplasty using the Mako robotic arm system.
  "Participants" throughout this posting is equivalent to the number of knees.
Period: Overall Study
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Started | 100
Completed | 89
Not Completed | 11
Not completed — Exclusion due to implant size | 5
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- Robotic Assisted Total Knee Arthroplasty: Participants who underwent primary total knee arthroplasty using the Mako robotic arm system.
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.78 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Intra-Operative Complications
Description: Surgeon assessment of standardized TKA complications (Healey et al. CORR 2012) both intra-operatively and at short term follow up. The nine complications relating to soft tissue damage for primary TKA that were assessed as part of this study were as follows: Blood loss, Vascular injury, MCL injury, Periprosthetic fracture, Extensor mechanism disruption, Patellofemoral dislocation, Tibiofemoral dislocation, Neurological impairment, Instability.
Time Frame: Subject will be assessed for these complications intra-operatively. The assessment occurs after the surgeon has completed the surgical procedure, but while the subject is still in the operating room with the surgeon.
Population: participants = knees.
Measure: Number; unit: intra-operative complications
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 89
intra-operative complications | 0

2. Primary Outcome: Intra-Operative Complications
Description: as for outcome 1
Time Frame: Subjects will be assessed for incidence of intra-operative complications at the conclusion of their hospital stay, or an average of 3 days post-operatively.
Population: participants = knees.
Measure: Number; unit: intra-operative complications
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 89
intra-operative complications | 0

3. Primary Outcome: Intra-Operative Complications
Description: as for outcome 1
Time Frame: 3 Month Post Op
Population: participants = knees.
Measure: Number; unit: intra-operative complications
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 89
intra-operative complications | 0
Statistical Analysis 1: Comparison: Robotic Assisted Total Knee Arthroplasty; Test type: Non-Inferiority or Equivalence — The Alternative Hypothesis: The Investigational Device (RIO) true event rate is non-inferior to 0.066 (event rate for manual TKA) with a non-inferiority margin of 0.06. The 0.066 rate is based on literature and 0.06 was determined in consultation with FDA; Rare Adverse Event Rate = 0, 95% CI 1-sided [upper limit 0.0331] — If the upper bound is <0.126 then the primary composite safety endpoint is met. After the surgeon completed the procedure, at the conclusion of the participant's hospital stay, and 3 months post-operative were used in this single analysis

4. Secondary Outcome: Change in the Radiographic Assessment of Limb Alignment From Pre-Operative to 3 Months Post-Operative
Description: Radiographic limb alignment of the operative knee according to the technique defined by Barrack et al. was assessed at the 3 month post-operative follow-up by two independent reviewers. The measured post-operative limb alignment was to be compared to the planned pre-operative limb alignment as extracted from the system log file.
Time Frame: pre-op plan, 3 Month Post Op
Population: Of the 89 patients who received a robotic assisted total knee arthroplasty as part of the IDE, 2 patients were excluded from analysis for the Secondary Endpoint only due to issues related to the accurate measurement of limb alignment from the radiographs available (not for reasons involving the surgical procedure or clinical outcomes).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 87
degrees | 1.54 (1.01)

5. Secondary Outcome: Participants With Limb Alignment Difference <4.38 Degrees
Description: The difference between the actual 3 month limb alignment was compared to the pre-op planned alignment. Any measurement difference <4.38 was considered a success; >4.38 degrees was considered a failure.
Time Frame: Pre-op Plan, 3 Month Post Op
Population: Participants = knees
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 87
Participants | 87
Statistical Analysis 1: Comparison: Robotic Assisted Total Knee Arthroplasty; Test type: Other — The analysis was performed using standard OC curves generated using Sample Size Analyzer® version 2.0 by Taylor Enterprise Inc. (Dr. Wayne A. Taylor); Alignment Difference <4.38 Degrees = 1, 95% CI 1-sided [lower limit 0.966] — Estimation Parameter is: proportion of participants with limb alignment difference <4.38 degrees If the lower bound is >0.95 then the assessment passes

6. Other Pre Specified Outcome: Patient Satisfaction - Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC)
Description: The WOMAC collects information specific to osteoarthritis outcomes. The patient-response questionnaire uses a visual analog scale for pain, measuring factors of general pain, stiffness, and function. Each question is scored from 0 to 4 for each set of factors, with 0 indicating no pain, stiffness, or limit in function, and 4 indicating extreme pain, stiffness, or limit in function. Total WOMAC scores range from 0 to 96 with lower values representing better outcomes.
  The posted mean, noted as a negative number, represents the mean DECREASE in total WOMAC score from pre-operative to 3 month post-operative patient assessment.
Time Frame: Pre-Op, 3 Month Post Op [change assessed between the two time periods]
Population: participants = knees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Number analyzed (Participants) | 89
units on a scale | -33.1 (20.04)
Statistical Analysis 1: Comparison: Robotic Assisted Total Knee Arthroplasty; Change from pre-op to 3 months; Test type: Non-Inferiority — The upper bound for the one-sided 95% confidence interval will be compared with -9. If the upper bound is less than -9, then non-inferiority holds; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -33.1, 95% CI 1-sided [upper limit -29.6] — If the upper bound is less than -9, then non-inferiority holds

ADVERSE EVENTS:
Time Frame: Subject enrollment to end of study.
Description: Participants = knees
Groups:
- Robotic Assisted Total Knee Arthroplasty: Participants who underwent primary total knee arthroplasty using the Mako robotic arm system.
  Note regarding serious AEs:
  Adhesions and arthrofibrosis are surgical complications that can result from knee surgery and present as stiffness and restriction of ROM. Reasons for stiffness and restriction of ROM after TKA are multifactorial and may be influenced by factors such as the patient's overall health, motivation, and compliance to their rehabilitation regimen. The Principal Investigator and study Investigators stated these adverse events are not related to the use of the Investigational Device.
Arm/Group | Robotic Assisted Total Knee Arthroplasty
Serious Adverse Events (participants affected / at risk) | 9/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic Assisted Total Knee Arthroplasty (N=100)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 4
Adhesions (Musculoskeletal and connective tissue disorders) | 4
Pulmonary Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days